CLINICAL TRIAL: NCT07163416
Title: Project for the Construction of the Italian Migraine Registry I-GRAINE-New
Brief Title: (Italian Migraine Registry, I-GRAINE-NEW)
Acronym: I-GRAINE-NEW
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 20/16
Record Dates: First submitted 2025-07-18; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Migraine Disorders
Keywords: Migraine,Register,Italy
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale Understanding the mechanisms and evolution of migraine is hampered by its nature as a chronic "evolutionary" condition. Patients often come to migraine centers after years of disabling disease, non-specific diagnoses and ineffective treatments. When patients are admitted to the center is therefore the time when their history in terms of disease evolution and healthcare costs is most effectively collected, but also when it is assumed that the treatment strategy offered to the patient will have a greater impact.

For this reason, it was decided to conduct a large-scale retrospective and prospective observational study in order to draw a detailed picture of the situation of patients not followed by a specialized center and of the natural history of the disease once the pathway at the specialized center has started.

Design A multicenter, observational, retrospective and prospective cohort study, aimed at obtaining a more detailed picture of the situation of patients not followed by a specialized center and of the natural history of the disease once the pathway at the specialized center has started.6,000 of the incident patients (defined as those who had their first visit during the 6 months preceding enrollment in the registry), will be invited to take part in a follow-up and expanded data collection study.

Patients will be consecutively enrolled by specialists at each individual site.. Eligible patients who agree to take part in the study by signing an informed consent form will be assessed clinically and through a direct interview with a structured questionnaire organized in several ad hoc sections.

Objectives: The aim of the study is:

analyze episodic and chronic migraine in Italy from an epidemiological point of view, especially in terms of prevalence of the two forms of migraine and their endophenotypes in different population subgroups; 2. characterize the demographic distribution and clinical characteristics of patients (including the definition of endophenotypes); 3. measure the influence of the disease on the patient's daily activity, in terms of disability (assessed using the validated MIDAS and HIT-6 scales); 4. study the clinical and care pathway (patient journey) and identify the preferred care pathways based on the characteristics of the patients and the migraine subtype; 5. evaluate the prescribed pharmacological treatments, medical visits and diagnostic procedures performed (ascertaining the degree of adherence to current guidelines); 6. analyze the use of health resources by migraine patients, with particular attention to their impact on the SNS.

Visits and Treatments:

Baseline Visit: Patients enrolled in the study will undergo a thorough clinical and neurological examination.

Follow-up Visits: Clinical data will continue to be collected over time, at each scheduled clinic visit based on the needs of clinical practice.

Study Population: Adult patients of both sexes with episodic or chronic migraine who have recently attended a specialized migraine center in the I-GRAINE-NEW registry.

Estimated Study Duration: The duration of each patient's participation in the study is 24 months from the date of the initial visit to the participating migraine site

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients(Age ≥ 18 years) of both sexes
* Diagnosis confirmed of episodic migraine ( <15 days/month ) with or without aura or chronic migraine (>15days/month) ,with or without headeche due to overuse of analgesics;
* Provision of signed and dated the Informed Consent Form before the inclusion in the study

Exclusion Criteria:

* Patients affected by other forms of primary or secondary headaches or in whom the diagnosis is not certain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The reference population for the registry IGRAINE includes adult patients of both sexes, suffering from episodic or chronic migraine, undergoing treatment at a specialized headache center.
  At the time of its launch, 46 headache centers distributed throughout Italy will participate in the registry. To ensure its representativeness, the study sample includes 10% of the total number of patients followed at the centers, selected randomly.
  The registry will be enrolled using the "systematic random" method. Participation in the study will be offered to the first patient at the first visit (incident patient) and to the first patient at the follow-up visit (prevalent patient) of each outpatient day at the clinical center.
  If the first patient in each category refuses, participation in the study will be offered to the next patient in order of visit in the same category (prevalent or incident). Researchers are advised NOT to skip patients so as not to create a selection bias in the population.
Sampling Method: Probability Sample
Enrollment: 2030 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Better definition of the dimensions of the migraine phenomenon in Italian headache centers | "Baseline visit or (day 1)"" through study completion, an average of 2 year"
  More appropriate estimate of the prevalence of migraines refractory to treatments.
  In particular:
  1.Identification of clinical endophenotypes that can be predictive of evolution and pharmacological .
  Allodynia will be assessed through the ASC 12 scale.
  1. Disability measured using the validated clinical scales MIDAS, HIT-6.
  2. Treatments for migraine attacks and preventive therapies
Information on the patient's level of awareness and knowledge of the migraine problem | Baseline visit ,through study completion, an average of 2year
  1. Information on the times and methods of access to treatments:
  1. evaluation of the interval between the onset of the pathology and access to medical care;
  2. health tourism (migration of patients to regions other than their own). 5. Critical issues of the current clinical governance and determination of the use of healthcare resources, and in particular:
  a. Presence or absence of regional PDTA b. Degree of adherence to diagnostic-therapeutic guidelines c. Proper or improper use of diagnostic tests d. Patient traceability e. Definition of the percentage of patients who access visits, tests and treatments through the NHS.

CONTACTS AND LOCATIONS:
Locations (1):
- Head, Irccs San Raffaele Roma S.r.l. - Unità per la cura e la ricerca su cefalee e dolore - Dipartimento di Neurologia, Via di Val di Cannuta 250, 00166 Roma (RM) - Italy, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No